CLINICAL TRIAL: NCT00399217
Title: Acute Intra-operative Testing of Subcutaneous Implantable Defibrillator Emulator and Parasternal Electrode, Acutely Implanted, for Comparison With Transvenous System
Brief Title: Further Acute Research of a Subcutaneous Implantable Defibrillator (S-ICD) System
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: DN-05290
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2010-05

CONDITIONS: Ventricular Fibrillation; Ventricular Tachycardia
Keywords: subcutaneous ICD; ICD; DFT; Pacing threshold; Polarity
MeSH Terms: conditions — Ventricular Fibrillation; Tachycardia, Ventricular | interventions — Drug Delivery Systems

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: Subcutaneous Implantable Defibrillator (S-ICD) system
Device: ICD

SUMMARY:
The purpose is to further evaluate the operation, safety, and feasibility of a subcutaneous implantable defibrillator (S-ICD) system in patients who require an implantable cardioverter defibrillator (ICD)for treating ventricular tachyarrhythmias. The S-ICD electrode and pulse generator emulator will be briefly implanted and tested during the standard implantation procedure of an ICD, but then the S-ICD system will be removed entirely.

DETAILED DESCRIPTION:
The objectives of this study are to further evaluate the S-ICD system's ability to identify and terminate induced ventricular tachyarrhythmias in patients acutely with an S-ICD emulator and parasternal electrode during the implant procedure of a standard transvenous ICD.

The active emulator is not a powered medical device and all elements of the test system are removed following the testing.

This acute intra-operative protocol will test the ability of the electrode and emulator to appropriately convert the arrhythmia and allos an assessment of post shock pacing.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring ICD therapy according to National Centre for Clinical Excellence (NICE) criteria are eligible
* And patients who require replacement of an existing transvenous ICD system are eligible

Exclusion Criteria:

* Patients unable or unwilling to provide informed consent
* Any conditions which precludes the subject's ability to comply with the study requirements, including completion of the study
* Females who are pregnant or lactating and pre-menopausal women who are unwilling to use adequate birth control for the duration of the study
* Participation in another investigational device trial at any time during the conduct of this study
* Patients with a serious medical condition and life expectancy of less than one year
* Patients with documented spontaneous and frequently recurring VT that is reliably terminated with anti-tachycardia pacing
* Patients with existing epicardial patches or subcutaneous electrodes in the left thoracic quadrant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients requiring ICD therapy
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2006-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Grace, MD, PhD, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital NHS Trust, Papworth Everard, Cambridge, United Kingdom

REFERENCES:
- [Derived] Bardy GH, Smith WM, Hood MA, Crozier IG, Melton IC, Jordaens L, Theuns D, Park RE, Wright DJ, Connelly DT, Fynn SP, Murgatroyd FD, Sperzel J, Neuzner J, Spitzer SG, Ardashev AV, Oduro A, Boersma L, Maass AH, Van Gelder IC, Wilde AA, van Dessel PF, Knops RE, Barr CS, Lupo P, Cappato R, Grace AA. An entirely subcutaneous implantable cardioverter-defibrillator. N Engl J Med. 2010 Jul 1;363(1):36-44. doi: 10.1056/NEJMoa0909545. Epub 2010 May 12. PMID 20463331